CLINICAL TRIAL: NCT06145282
Title: Non-myeloablative Phase I/II Haploidentical HCT Study for Patients With Sickle Cell Disease, Including Compromised Organ Function
Brief Title: Non-myeloablative Haploidentical HCT Study for Patients With Sickle Cell Disease, Including Compromised Organ Function
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10001635; 001635-H
Record Dates: First submitted 2023-11-22; First posted 2023-11-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12-17

CONDITIONS: Sickle Cell Disease
Keywords: Organ Damage; Hematopoietic Cell Transplant; Haploidentical; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Abatacept

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): All participants will receive the same dose of the investigational briquilimab antibody and abatacept added to the NIH-established regimen of alemtuzumab-TBI-sirolimus and infusion of filgrastim-mobilized peripheral blood hematopoietic cells from haploidentical related donors. Cohort 1 will receive a single dose of PT-Cy; 50 mg/kg, on day +3 post-HCT
  Interventions: Drug: Non-myeloablative haploidentical peripheral blood stem cell transplantation with briquilimab and abatacept
- Cohort 2 (Experimental): All participants will receive the same dose of the investigational briquilimab antibody and abatacept added to the NIH-established regimen of alemtuzumab-TBI-sirolimus and infusion of filgrastim-mobilized peripheral blood hematopoietic cells from haploidentical related donors. Cohort 2 will receive a total of two doses of PT-Cy; 50mg/kg, on days +3 and +4 (total 100 mg/kg) post-HCT
  Interventions: Drug: Non-myeloablative haploidentical peripheral blood stem cell transplantation with briquilimab and abatacept

INTERVENTIONS:
Drug: Non-myeloablative haploidentical peripheral blood stem cell transplantation with briquilimab and abatacept — All participants will receive the same dose of the investigational briquilimab antibody and abatacept added to the NIH-established regimen of alemtuzumab-TBI-sirolimus and infusion of filgrastim-mobilized peripheral blood hematopoietic cells from haploidentical related donors.

SUMMARY:
Background:

Sickle cell disease (SCD) is a genetic disorder where red blood cells, that carry oxygen, are stiff and become stuck in small blood vessels. As a result, affected patients can experience severe pain and serious organ damage. SCD can be cured with a hematopoietic cell transplant (HCT), that is, when they receive blood stem cells from a family donor. But HCT can also have serious side effects, especially in people with organ damage. Researchers want to find ways to make HCT safer for everyone.

Objective:

To test a new combination of drugs (briquilimab, abatacept, and alemtuzumab), used along with radiation, in people undergoing HCT for SCD.

Eligibility:

People aged 16 and older with SCD. They must be eligible for HCT and have a family member who is a good donor match. Donors must be aged 4 and older.

Design:

Participants with SCD will be screened. They will have blood tests and tests of organs including their heart and lung function. Donors will have blood drawn.

Participants with SCD will have a tube inserted into a blood vessel in their chest (intravenously). This line will remain in place up to 2 months; it will be used to draw blood and administer the donor cells and other medications.

Briquilimab will be administered intravenously 1 time, along with other drugs used to prepare for HCT. Participants will receive abatacept 6 times, from just before they receive their donor cells until 6 months after. Participants will undergo radiation therapy and take other drugs that are standard for HCT. Most HCT recipients remain in the hospital for about 30 days after HCT.

Follow-up visits will continue for 5 years....

DETAILED DESCRIPTION:
Study Description:

Haploidentical hematopoietic cell transplantation offers a widely available curative option for individuals with sickle cell disease. The goal is to reverse SCD while avoiding unacceptable graft rejection, graft-versus-host disease, infectious complications, and hyperinflammatory responses. We hypothesize that a moderate amount of immunosuppression will maximize efficacy while avoiding unacceptable toxicity.

Objectives:

Primary Objective:

-Evaluate the regimen success rate where success is defined as successful engraftment (persistent donor chimerism and free of acute SCD complications) and absence of acute grade 3 or higher GVHD or moderate to severe chronic GVHD evaluated at 1 year posttransplant.

Secondary Objectives:

* Event-free survival and overall survival.
* Incidence of recipient-type hemoglobin defined as HbS >10% when donors have HbAA and HbS >50% when donors have sickle cell trait (HbAS).
* The proportion of patients with myeloid chimerism >= 95% at 1 and 2 years post-HCT.
* Incidence of acute and chronic GVHD.
* Prevalence of donor type hemoglobin at 1-year post-transplant in SCD patients who have not been transfused in the previous 3 months.
* Incidence of viral reactivation and disease.
* Incidence of autoimmune and hyperinflammatory complications.
* Incidence of hematologic malignancies.
* Transplant-related mortality.

Exploratory Objective:

* Perform gene therapy research involving cell culture or genetic manipulation to produce normal or therapeutic hemoglobin on excess autologous CD34+ cells collected from recipients.
* Evaluate the impact of this non-myeloablative conditioning regimen on organs including the heart, lung, kidneys, liver, brain, neurocognitive function, and endocrine organs
* Evaluate the impact of this non-myeloablative conditioning regimen on quality of life.

Endpoints:

Primary Endpoint:

-The percentage of SCD patients at 1 year (+/- 3 months) posttransplant who have not experienced graft failure and who are without severe graft-versus-host disease (defined as grade 3 and higher acute GVHD and moderate to severe chronic GVHD).

Secondary Endpoints:

* Total hemoglobin and percent HbS levels
* Percent donor myeloid chimerism and donor CD3 chimerism
* Day of neutrophil engraftment
* Day of platelet engraftment
* RBC transfusion requirement
* Rates of acute and chronic GVHD
* Rates of viral reactivation and disease
* Rates of autoimmune and hyperinflammatory complications
* Transplant-related mortality
* Non-transplant-related mortality
* Rates of graft failure
* Rates of leukemia and related disorders

Exploratory Endpoint:

Completion of gene therapy research involving cell culture or genetic manipulation to produce normal or therapeutic hemoglobin on excess autologous CD34+ cells collected from recipients.

Organ function and quality of life

ELIGIBILITY:
* INCLUSION CRITERIA:

Recipient:

Participants must fulfill one disease category, either at least one organ damage or no other access to curative therapy.

1. Adult patients with sickle cell disease at high risk for disease-related morbidity or mortality, according to A, B, C, D, or E or complication(s) not ameliorated by SICKLE CELL-SPECIFC THERAPIES (F):

   A. Stroke defined as a clinically significant neurologic event that is accompanied by an infarct on cerebral MRI OR an abnormal trans-cranial Doppler examination (>=200 m/s); OR

   B. Silent cerebral infarct defined as an infarct-like lesion based on an MRI signal abnormality at least 3 mm in one dimension and visible in two planes on FLAIR or T2- weighted images (or similar image with 3D imaging) and documented neurological examination performed by a neurologist demonstrating the participant has a normal neurologic examination or an abnormality on examination that could not be explained by the location of the brain lesion(s); OR

   C. Sickle cell-related renal insufficiency defined by a creatinine level >=1.5 times the upper limit of normal and kidney biopsy consistent with sickle cell nephropathy OR nephrotic syndrome; OR

   D. Tricuspid regurgitant jet velocity (TRV) of >=2.5 m/s at least 3 weeks after a vaso-occlusive crisis and/or right heart catheterization-documented pulmonary hypertension; OR

   E. Sickle hepatopathy defined as EITHER ferritin >1000 mcg/L OR direct bilirubin >0.4 mg/dL at baseline AND a platelet count <250 K/microliter (without vaso-occlusive crisis); OR

   F. Any one of the below complications:

   Complication: Vaso-occlusive crises; Eligible for HCT: >1 hospital admission per year while on a therapeutic dose of a SCD treatment/medication

   Complication: Acute chest syndrome (ACS); Eligible for HCT: Any ACS while on SCD treatment/medication

   Pediatric patients with sickle cell disease at high risk for disease-related morbidity or mortality, defined as A, B, C, D, E, or F

   A. A neurological event resulting in focal neurologic deficits that lasted >= 24 hours (classical clinical definition of stroke, not requiring imaging studies of the brain) OR a focal neurological event resulting in abnormalities on T2-weighted or FLAIR images using a MRI scan, indicative of an acute infarct, with no other reasonable medical explanation (definition of a stroke supported with MRI imaging scans of the brain), OR both; OR

   B. Abnormal transcranial Doppler (TCD) measurement with a timed average maximum mean velocity of at least 200 cm/sec in the terminal portion of the internal carotid or proximal portion of middle cerebral artery or if the imaging TCD method is used > 185 cm/sec plus evidence of intracranial vasculopathy; OR

   C. Silent Cerebral Infarct defined as an infarct-like lesion based on an MRI signal abnormality at least 3 mm in one dimension and visible in two planes on FLAIR or T2-weighted images (or similar image with 3D imaging) and documented neurological examination performed by a neurologist demonstrating the participant has a normal neurologic examination or an abnormality on examination that could not be explained by the location of the brain lesion(s); OR

   D. Three acute severe vaso-occlusive pain episodes requiring hospitalization and recalcitrant to maximum medical therapy; OR

   E. At least one acute chest syndrome episode resulting in intensive care admission requiring nonmechanical ventilatory support: simple nasal cannula, face mask that requires oxygen content (venti mask, non-rebreather), simple nasal cannula, face mask oxygen (e.g. ventimask, nonrebreather), continuous positive airway pressure, synchronized inspiratory positive airway pressure, bilevel positive airway pressure, high flow nasal cannula or invasive mechanical ventilatory support (delivered by endotracheal tube or tracheostomy); OR

   F. Right heart catheterization confirmed pulmonary hypertension defined as pulmonary artery pressure >25 mmHg
2. AND evidence of severe organ damage with at least one of the following who are typically excluded from other HCT protocols:

   A. Kidney damage: CrCl <60 mL/min/1.73m^2 cystatin C-based or iothalamate/iohexol-based or other equivalent GFR testing including patients on hemodialysis or peritoneal dialysis

   B. Heart damage: Ejection fraction 35-40%

   C. Liver damage: Bridging fibrosis, cirrhosis, direct bilirubin >= 2x the upper limit of normal and/or ALT >= 5x the upper limit of normal

   D. Lung damage: Adjusted diffusion capacity of carbon monoxide (DLCO) 35-40% OR who have no other option for curative therapy (including allogeneic HCT, gene therapy, or gene editing studies) on a different SCD HCT protocol.
3. Non disease-specific:

   * Male or female, age >=18 years (pediatric subjects >=16 years may be enrolled after 6 successful adult transplants)
   * Haploidentical relative donor available
   * Ability to comprehend and willing to sign an informed consent before the initiation of any study procedures
   * Negative serum or urine b-HCG, when applicable
   * Agree to use birth control for 12 months after drug product infusion.

     * Female subjects must agree to use a medically acceptable method of birth control such as an oral contraceptive, intrauterine device, barrier and spermicide, or contraceptive implant/injection from start of screening through 12 months after drug product infusion.
     * Male subjects must agree to use effective contraception (including condoms) from start of screening through 12 months after drug product infusion.
   * Stated willingness to comply with all study procedures and availability for the duration of the study

Donor:

Haploidentical relative donor deemed suitable and willing to donate, per clinical evaluations. Donors age 4 or older and >=20 kg, eligible to donate hematopoietic stem cells, and who are additionally willing to donate blood for research. Related donors will be evaluated in accordance with existing Standard NIH Policies and Procedures for determination of eligibility and suitability for clinical donation. Note that participation in this study is offered to all related donors, but is not required for a donor to make a stem cell donation, so it is possible that not all related donors will enroll onto this study.

EXCLUSION CRITERIA:

Recipient:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Available HLA-matched sibling donor
* ECOG performance status of 3 or more.
* DLCO <35% predicted (corrected for hemoglobin).
* Baseline oxygen saturation of <85% or PaO2 <70 mmHg
* Left ventricular ejection fraction: <35% estimated by ECHO
* Evidence of uncontrolled bacterial, viral, or fungal infections (currently taking medication and progression of clinical symptoms) within one month prior to starting the conditioning regimen. HCT candidates with pre-transplant respiratory viral infections will undergo careful clinical assessment with the help of our transplant infectious disease team for lower respiratory tract disease, which may include thorough physical examination, imaging, and/or bronchoalveolar lavage. In case of lower respiratory tract disease or severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) positivity, the transplant will be delayed until resolution.
* Major anticipated illness or organ failure incompatible with survival from PBSC transplant.
* Pregnant or breastfeeding
* Donor specific anti-HLA antibodies (DSAs) >=2000 Mean Fluorescence Intensity (MFI)
* Patients seronegative for EBV who have EBV seropositive donors

Ages: 4 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-12-28 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2027-11-26 (Estimated)

PRIMARY OUTCOMES:
Evaluate the regimen success rate where success defined as successful engraftment and absence of acute grade 3 or higher GVHD or moderate to severe chronic GVHD evaluated at 1 yr post-transplant | 1 year (+/- 3 months)
  The percentage of SCD patients at 1 year (+/- 3 months) post-transplant who have not experienced graft failure and who are without severe graft-versus-host disease (defined as grade 3 and higher acute GVHD and moderate to severe chronic GVHD).

SECONDARY OUTCOMES:
Event-free survival and overall survival | length of study
Viral reactivation and disease | length of study
Autoimmune and hyperinflammatory complications | length of study

CONTACTS AND LOCATIONS:
Overall Officials: Courtney F Joseph, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001635-H.html

DOCUMENTS (1):
  • Informed Consent Form (2024-11-07): https://cdn.clinicaltrials.gov/large-docs/82/NCT06145282/ICF_000.pdf